CLINICAL TRIAL: NCT04348474
Title: Open Label, Multicentric, Non Randomized, Exploratory Clinical Trial to Assess the Efficacy and Safety of Hydroxychloroquine and Azithromycin for the Treatment of Mild Acute Respiratory Syndrome (COVID-19) Caused by SARS-CoV-2 Virus
Brief Title: Efficacy and Safety of Hydroxychloroquine and Azithromycin for the Treatment of Ambulatory Patients With Mild COVID-19
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Azidus, the CRO hired for this study by Prevent Senior has lost the interest to conduct this study.
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIAPRE0420OR
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCQ + AZT (Experimental): All patients included in the study will receive hydroxychloroquine (HCQ) 400 mg (00 mg BID on D1 and 400 mg/day on D2 to D7) and azithromycin (AZT) (500 mg/ 5 days) on top of standard care.
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Azithromycin Tablets

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — All patients included in the study will receive HCQ (400 mg BID on D1 and 400 mg/day on D2 to D7) for 7 days.
  Other Names: Reuquinol
Drug: Azithromycin Tablets — All patients included in the study will receive AZT 500 mg per day for 5 days.
  Other Names: Azithromycin

SUMMARY:
This is an exploratory study to evaluate the efficacy of hydroxychloroquine (400 mg BID on D1 and 400 mg/day on D2 to D7) and azithromycin (500 mg/ 5 days) to treat mild ambulatory COVID-19 patients.

DETAILED DESCRIPTION:
This is an exploratory study to evaluate the efficacy of hydroxychloroquine (400 mg BID on D1 and 400 mg/day on D2 to D7) and azithromycin (500 mg/ 5 days) to treat mild ambulatory COVID-19 patients.

We aim to demonstrate decrease in hospital related complications among ambulatory patients with mild COVID-19 by treating them with HCQ and AZT on top of standard care compared to patients who receive standard care only.

Ambulatory patients on day 3 of symptoms and with confirmed diagnosis of COVID-19 will receive the treatment.

Patients that do not fulfill the inclusion/exclusion criteria or that is not willing to participate in the study will be invited to consent the use of their data as part of a "control" group.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from patient or legal representative.
2. Male or female, and:

   1. aged ≥ 70 years; or
   2. aged < 70 with associated risk factors (chronic obstructive pulmonary disease; heart failure, immunosuppressed, obesity (BMI ≥ 35) uncontrolled diabetes and uncontrolled systemic arterial hypertension)
3. One or more mild symptoms characteristic of COVID-19 for 3 days, such as fever, cough and signs of respiratory distress, which do not require hospitalization.

Exclusion Criteria:

1. Participating in another RCT in the past 12 months;
2. Known allergy to HCQ or chloroquine
3. Any contraindication to HTC or AZT, including retinopathy and prolonged QT,
4. Severely reduced LV function
5. Severely reduced renal function;
6. Pregnancy or breast feeding
7. Any other clinical condition which, in the opinion of the principal investigator, would not allow safe completion of the protocol and safe administration of the investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Condition | 28 days
  Ordinal scale (7 points ordinal scale that measures illness severity over time)

SECONDARY OUTCOMES:
Hospitalization | 28 days
  Number of patients that needed to be hospitalized
Change in Clinical Condition | 28 days
  Time for normalization of body temperature
Change in Clinical Condition | 28 days
  Time for normalization of of respiratory rate
Change in Clinical Condition | 28 days
  Time for cough relief
Rate of mortality within 28-days | 28 days
  Evaluation of change in acute respiratory syndrome
Change in Clinical Condition related to comorbidity | 28 days
  Subgroup analysis by comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Prevent Senior Private Operadora de Saúde LTDA., São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.